CLINICAL TRIAL: NCT07005674
Title: Effectiveness and Cost-effectiveness of a Community-based Nine-week Multi-component Group-based Cycling Intervention Versus a Single Cycle Training Session to Increase Cycling Participation: the Cycle Nation Communities Randomised Controlled Trial
Brief Title: Cycle Nation Communities: Increasing Cycling in Glasgow
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Professor Jason Gill, Professor, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 200240325; NE/W005042/1 (Other Grant/Funding Number: Natural Environment Research Council)
Record Dates: First submitted 2025-05-22; First posted 2025-06-05 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: Cycling; Bicycle; Communities; Randomised controlled trial

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with two groups, Cycle Nation programme and Cycling Scotland single standard cycling session
Who Masked: Outcomes Assessor
Masking Description: Members of the research team that perform measurements are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycle Nation intervention (Experimental)
  Interventions: Behavioral: Cycle Nation
- Cycling Scotland standard cycling session (Active Comparator)
  Interventions: Behavioral: Cycling Scotland standard cycling session

INTERVENTIONS:
Behavioral: Cycle Nation — Participants will be asked to attend nine weekly 90-minute face-to-face sessions, delivered by trained facilitators at community cycling organisations. Sessions include off road cycling skills and on-road group rides, behaviour change techniques (e.g. goal setting), and bicycle maintenance training. Two extra group rides will be offered during the programme for additional practice, along with two catch-up sessions at the end for those who missed any content. Participants will be added to a WhatsApp group to encourage peer communication. Bicycles, helmets, and locks will be loaned to participants for 10-12 weeks to support participation.
  Arms: Cycle Nation intervention
Behavioral: Cycling Scotland standard cycling session — Participants will be asked to participate in Cycling Scotland's 'Introduction to On-Road Cycling' a single 2-2.5-hour session that is offered as standard. The session covers key cycling skills such as hazard awareness, road positioning, and communicating with other road users. Activities are tailored to participants' needs and may include navigating junctions, using shared infrastructure, and performing U-turns. Bicycles and helmets will be provided for the session.
  Arms: Cycling Scotland standard cycling session

SUMMARY:
This randomised controlled trial will evaluate the effects of a 9-week multi-component group-based cycling programme (Cycle Nation) versus a standard single cycle training session on self-reported cycling, health and wellbeing outcomes. Participants are adults that do not regularly cycle, who will be randomly allocated to each arm of the study. Outcomes will be assessed at baseline, post-programme, and at 12 months from baseline. Cost effectiveness will be assessed, and a process evaluation will be conducted.

DETAILED DESCRIPTION:
Cycling improves physical and mental health, lowering risks of major diseases and reducing stress while enhancing wellbeing and fitness. It is a time-efficient way to increase physical activity and, when replacing motorised transport, reduces air pollution, carbon emissions, and traffic congestion. However, cycling participation in the UK remains low; only 10% of adults cycle at least weekly. This is a missed opportunity to enhance population health, lower health service costs, reduce environmental impact, and improve health related quality of life. Evidence suggests that over 50% of UK adults are interested in cycling more, therefore the potential to increase cycling is substantial.

Non-cyclists report numerous barriers, spanning the individual, social, and environmental factors of the socio-ecological model. While improvements to cycling infrastructure can address some environmental barriers, they alone are insufficient to drive substantial increases in cycling. While many organisations offer standard single or short-term cycling sessions, these often address isolated components rather than taking an integrated approach. In contrast, Cycle Nation is an integrated group-based 9-week multi-component intervention, targeting multiple individual and social barriers over a sustained period to maximise effectiveness.

Initially co-developed and piloted in collaboration with British Cycling and HSBC-UK as a workplace programme for employees, it has since been adapted for community settings in Manchester and Glasgow. Findings of these studies have demonstrated feasibility, acceptability, and short-term effectiveness. However, Cycle Nation has not yet been rigorously tested in a powered randomised controlled trial (RCT), nor had its long-term effectiveness or cost-effectiveness evaluated.

This is a pragmatic, two-arm RCT to assess the effect of the Cycle Nation programme in comparison to a single cycling training session. The interventions will be delivered by community-based cycling delivery partners across Glasgow, UK, with up to six organisations delivering the Cycle Nation programme (intervention) and one delivering the standard single introduction to road cycling session offered by Cycling Scotland (comparison).

The primary objective is to evaluate the effect of the Cycle Nation programme versus a standard single session on the proportion of participants cycling at least weekly at 12 months. Secondary objectives are to a) to evaluate the effect of the Cycle Nation programme versus a standard cycling session on self-reported health and wellbeing at 12 months, b) to evaluate the within-trial cost-effectiveness of the Cycle Nation programme at 12 months (and longer pending within trial findings), c) to assess how (well) Cycle Nation is delivered and examine how the core causal mechanisms function, and d) to determine how contextual factors contribute to variations in outcome and engagement with the Cycle Nation intervention.

ELIGIBILITY:
Inclusion Criteria:

Can ride a bicycle Self-identified infrequent cyclists (currently cycle less than once per month) Aged 18 years or over Willing to provide informed consent Willing to partake in measurements Willing to be randomised to intervention or control arm Have a good understanding of the English language Not have a contraindication to moderate intensity physical activity as assessed by the adapted Physical Activity Readiness Questionnaire-Plus (PAR-Q+) Able to attend in-person sessions (at least 6 out of 9 sessions) Intend to still be in the UK by November 2026

Exclusion Criteria:

Cannot cycle (i.e. cannot balance and/or have never learnt to cycle) Frequent or regular cyclists (i.e. currently cycle at least once a month, confident riding on roads) Less than 18 years old Not willing to provide informed consent Not willing to partake in measurements Not willing to be randomised to the intervention or control arm Cannot speak basic English Have a contraindication to moderate intensity physical activity as assessed by the adapted Physical Activity Readiness Questionnaire-Plus (PAR-Q+) Not able to attend in-person sessions (less than 6 out of 9 sessions) Not intending to still be in the UK by November 2026

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants cycling (for any purpose) | From baseline to 12 months follow-up
  Change in number (proportion) of participants cycling (for any purpose) over past four weeks at 12 months

SECONDARY OUTCOMES:
Proportion of participants cycling (for any purpose) | From baseline to 12 weeks follow-up
  Change in number (proportion) of participants cycling (for any purpose) over past four weeks at 12-weeks follow-up
Number of cycling journeys (for any purpose) | From baseline to 12-weeks and 12-months follow-up
  Change in the number of cycling journeys (for any purpose) over past four weeks at 12 weeks and at 12 months follow-up
Number of cycling journeys (leisure) | From baseline to 12 weeks and 12 months follow-up
  Change in the number of cycling journeys (for leisure) over past four weeks at 12 weeks and at 12 months follow-up
Number of cycling journeys (commuting) | From baseline to 12 weeks and 12 months follow-up
  Change in the number of cycling journeys (for commuting) over past four weeks at 12 weeks and at 12 months follow-up
Number of cycling journeys (errands) | From baseline to 12 weeks and 12 months follow-up
  Change in the number of cycling journeys (for errands) over past four weeks at 12 weeks and at 12 months follow-up
Total duration of weekly cycling (for any purpose) | From baseline to 12 weeks and 12 months follow-up
  Change in total duration (minutes) of weekly cycling (for any purpose) over past four weeks at 12 weeks and at 12 months follow-up
Total duration of weekly cycling (leisure) | From baseline to 12 weeks and 12 months follow-up
  Change in total duration (minutes) of weekly cycling (for leisure) over past four weeks at 12 weeks and at 12 months follow-up
Total duration of weekly cycling (commuting) | From baseline to 12 weeks and 12 months follow-up
  Change in total duration (minutes) of weekly cycling (for commuting) over past four weeks at 12 weeks and at 12 months follow-up
Total duration of weekly cycling (errands) | From baseline to 12 weeks and 12 months follow-up
  Change in total duration (minutes) of weekly cycling (for errands) over past four weeks at 12 weeks and at 12 months follow-up
Number of private car journeys | From baseline to 12 weeks and 12 months follow-up
  Change in time of private car journeys over past four weeks at 12 weeks and at 12 months
Number of taxi journeys | From baseline to 12 weeks and 12 months follow-up
  Change in the number of taxi journeys over past four weeks at 12 weeks and at 12 months follow-up
Total duration of taxi journeys | From baseline to 12 weeks and 12 months follow-up
  Change in total duration (minutes) of weekly taxi journeys over past four weeks at 12-weeks and at 12 months follow-up
Number of public transport journeys | From baseline to 12 weeks and 12 months follow-up
  Change in the number of weekly public transport journeys over past four weeks at 12 weeks and at 12 months follow-up
Total duration of public transport journeys | From baseline to 12 weeks and 12 months follow-up
  Change in total duration (minutes) of weekly public transport journeys over past four weeks at 12-weeks and at 12 months
Number of walking journeys | From baseline to 12 weeks and 12 months follow-up
  Change in the number of walking journeys over past four weeks at 12 weeks and at 12 months
Total duration of walking journeys | From baseline to 12 weeks and 12 months follow-up
  Change in total duration (minutes) of walking journeys over past four weeks at 12-weeks and at 12 months
Perception of cycling safety | From baseline to 12 weeks and 12 months follow-up
  Change in perception of cycling safety at 12 weeks and 12 months follow-up
Perceptions of environment | From baseline to 12 weeks and 12 months follow-up
  Change in perception of environment at 12 weeks and 12 months follow-up
Confidence to cycle | From baseline to 12 weeks and 12 months follow-up
  Change in confidence to cycle at 12 weeks and 12 months
Motivation for cycling | From baseline to 12 weeks and 12 months follow-up
  Change in motivation (intrinsic motivation, identified regulation, introjected regulation, external regulation, and amotivation for exercise) using the Behavioural Regulation in Exercise Questionnaire (BREQ-2) at 12 weeks and 12 months
Self-esteem | From baseline to 12 weeks and 12 months follow-up
  Change in self-esteem (Rosenberg Self-Esteem Questionnaire) at 12 weeks and 12 months
Vitality | From baseline to 12 weeks and 12 months follow-up
  Change in vitality score (Subjective Vitality Scale) at 12 weeks and 12 months
Health related quality of life | From baseline to 12 weeks and 12 months follow-up
  Change in health-related quality of life score (EQ-5D-5 L) at 12 weeks and 12 months
Capability wellbeing | From baseline to 12 weeks and 12 months follow-up
  Change in capability wellbeing score (ICECAP-A) at 12 weeks and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gill, PhD, Principal Investigator — University of Glasgow; Cindy Gray, PhD, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
At the end of the project, anonymised/pseudonymised/de-identified research data will be deposited with the UK Data Service ReShare Repository.

REFERENCES:
- [Background] Connell H, Logan G, Somers C, Baker G, Broadfield S, Bunn C, Harper LD, Kelly P, McIntosh E, Pell JP, Puttnam J, Robson S, Gill JMR, Gray CM. Development and optimisation of a multi-component workplace intervention to increase cycling for the Cycle Nation Project. Front Sports Act Living. 2022 Oct 26;4:857554. doi: 10.3389/fspor.2022.857554. eCollection 2022. PMID 36385778
- [Background] Kelly P, Williamson C, Baker G, Davis A, Broadfield S, Coles A, Connell H, Logan G, Pell JP, Gray CM, Gill JM; Cycle Nation Project. Beyond cycle lanes and large-scale infrastructure: a scoping review of initiatives that groups and organisations can implement to promote cycling for the Cycle Nation Project. Br J Sports Med. 2020 Dec;54(23):1405-1415. doi: 10.1136/bjsports-2019-101447. Epub 2020 Apr 8. PMID 32269057